CLINICAL TRIAL: NCT05600426
Title: A Phase III Randomized Trial Comparing Unrelated Donor Bone Marrow Transplantation With Immune Suppressive Therapy for Newly Diagnosed Pediatric and Young Adult Patients With Severe Aplastic Anemia (TransIT, BMT CTN 2202)
Brief Title: A Trial Comparing Unrelated Donor BMT With IST for Pediatric and Young Adult Patients With Severe Aplastic Anemia (TransIT, BMT CTN 2202)
Acronym: TransIT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Center for International Blood and Marrow Transplant Research (Network); National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); North American Pediatric Aplastic Anemia Consortium (Unknown); Pediatric Transplantation and Cellular Therapy Consortium (Other); Blood and Marrow Transplant Clinical Trials Network (Network)
Responsible Party: Principal Investigator, David Williams, Chief - Division of Hematology/Oncology, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2020-0438; 1UG3HL157564-01A1 (NIH); 1U24HL157560-01A1 (NIH)
Record Dates: First submitted 2022-10-20; First posted 2022-10-31 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Severe Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — Cyclosporine; Antilymphocyte Serum; thymoglobulin; Methotrexate; fludarabine; Cyclophosphamide; Whole-Body Irradiation; Immunosuppression Therapy

STUDY DESIGN:
Intervention Model Description: Unblinded, stratified, multi-center, phase 3, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immunosuppressive Therapy (Active Comparator): Patient will receive standard immunosuppressive therapy combination of drugs: horse anti-thymocyte globulin (ATG) and cyclosporine.
  Interventions: Drug: cyclosporine; Drug: horse anti-thymocyte globulin (ATG); Procedure: Immunosuppressive Therapy (IST)
- Matched Unrelated Stem Cell Transplant (Active Comparator): Patient will under go matched unrelated donor transplant of hematopoietic stem cells as their therapy using fludarabine, cyclophosphamide, rabbit anti-thymocyte globulin (ATG), and low-dose total body irradiation (TBI) as preparative regimen and cyclosporine and methotrexate for graft versus host disease (GVHD) prevention.
  Interventions: Drug: cyclosporine; Procedure: Matched Unrelated Donor Hematopoetic Stem Cell Transplant; Drug: rabbit anti-thymocyte globulin (ATG); Drug: Methotrexate; Drug: Fludarabine; Drug: Cyclophosphamide; Radiation: low-dose total body irradiation (TBI)

INTERVENTIONS:
Drug: cyclosporine — cyclosporine
Procedure: Matched Unrelated Donor Hematopoetic Stem Cell Transplant — Matched Unrelated Donor (MUD) Hematopoietic Stem Cell Transplantation (HSCT)
  Arms: Matched Unrelated Stem Cell Transplant
Drug: horse anti-thymocyte globulin (ATG) — horse anti-thymocyte globulin (ATG)
  Other Names: ATGAM
  Arms: Immunosuppressive Therapy
Drug: rabbit anti-thymocyte globulin (ATG) — rabbit anti-thymocyte globulin (ATG)
  Other Names: thymoglobulin
  Arms: Matched Unrelated Stem Cell Transplant
Drug: Methotrexate — methotrexate
  Arms: Matched Unrelated Stem Cell Transplant
Drug: Fludarabine — fludarabine
  Arms: Matched Unrelated Stem Cell Transplant
Drug: Cyclophosphamide — cyclophosphamide
  Arms: Matched Unrelated Stem Cell Transplant
Radiation: low-dose total body irradiation (TBI) — low-dose total body irradiation (TBI)
  Arms: Matched Unrelated Stem Cell Transplant
Procedure: Immunosuppressive Therapy (IST) — Immunosuppressive Therapy (IST)
  Arms: Immunosuppressive Therapy

SUMMARY:
Severe Aplastic Anemia (SAA) is a rare condition in which the body stops producing enough new blood cells. SAA can be cured with immune suppressive therapy or a bone marrow transplant. Regular treatment for patients with aplastic anemia who have a matched sibling (brother or sister), or family donor is a bone marrow transplant. Patients without a matched family donor normally are treated with immune suppressive therapy (IST). Match unrelated donor (URD) bone marrow transplant (BMT) is used as a secondary treatment in patients who did not get better with IST, had their disease come back, or a new worse disease replaced it (like leukemia).

This trial will compare time from randomization to failure of treatment or death from any cause of IST versus URD BMT when used as initial therapy to treat SAA.

The trial will also assess whether health-related quality of life and early markers of fertility differ between those randomized to URD BMT or IST, as well as assess the presence of marrow failure-related genes and presence of gene mutations associated with MDS or leukemia and the change in gene signatures after treatment in both study arms.

This study treatment does not include any investigational drugs. The medicines and procedures in this study are standard for treatment of SAA.

DETAILED DESCRIPTION:
This study is a multi-center randomized phase III trial to compare the failure free survival between those randomized to IST vs 9-10/10 HLA matched URD BMT. The study will also address patient-reported outcomes and gonadal function in each arm and explore critical biological correlates including assessing germline genetic mutations associated with pediatric SAA that may lead to a predisposition to the disease and the risk of development of clonal hematopoiesis following IST vs BMT in pediatric and young adult SAA.

This clinical trial will randomize 234 children/AYA over 3.3-4.7 years at a 1:1 ratio between initial treatment with immune suppression therapy (IST) with horse ATG (hATG)/cyclosporine (CsA) versus well- matched (9-10/10 allele) unrelated donor (URD) bone marrow transplantation (BMT) using a regimen of rabbit ATG (rATG)/fludarabine/cyclophosphamide and 200 cGy TBI. Duration of subject participation for all study procedures in this study will be up to 2 years after treatment; a single later timepoint between 3 and 5 years will be collected to follow patients for specific protocol defined late effects and survival.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in the randomized trial, an individual must meet all the following criteria:

1. Provision of signed and dated informed consent form for the randomized trial by patient and/or legal guardian.
2. Age ≤25 years old at time of randomized trial consent.
3. Confirmed diagnosis of idiopathic SAA, defined as:

   1. Bone marrow cellularity <25%, or <30% hematopoietic cells.
   2. Two of three of the following (in peripheral blood): neutrophils <0.5 x 10^9/L, platelets <20 x 10^9/L, absolute reticulocyte count <60 x 10^9/L or hemoglobin <8 g/dL.
4. No suitable fully matched related donor available (minimum 6/6 match for HLA-A and B at intermediate or high resolution and DRB1 at high resolution using DNA based typing).
5. At least 2 unrelated donors noted on NMDP search who are well matched (9/10 or 10/10 for HLA-A, B, C, DRB1, and DQB1 using high resolution).
6. In the treating physician's opinion, no obvious contraindications precluding them from BMT or IST.

Exclusion Criteria:

1. Presence of Inherited bone marrow failure syndromes (IBMFS). The diagnosis of Fanconi anemia must be excluded by diepoxybutane (DEB) or equivalent testing on peripheral blood or marrow. Telomere length testing should be sent on all patients to exclude Dyskeratosis Congenita (DC), but if results are delayed or unavailable and there are no clinical manifestations of DC, patients may enroll. If patients have clinical characteristics suspicious for Shwachman-Diamond syndrome, this disorder should be excluded by pancreatic isoamylase testing or gene mutation analysis (note: pancreatic isoamylase testing is not useful in children <3). Other testing per center may be performed to exclude IBMFS.
2. Clonal cytogenetic abnormalities or Fluorescence In-Situ Hybridization (FISH) pattern consistent with pre- myelodysplastic syndrome (pre-MDS) or MDS on marrow examination.
3. Known severe allergy to ATG.
4. Prior allogeneic or autologous stem cell transplant.
5. Prior solid organ transplant.
6. Infection with human immunodeficiency virus (HIV).
7. Active Hepatitis B or C. This only needs to be excluded in patients where there is clinical suspicion of hepatitis (e.g., elevated LFTs).
8. Female patients who are pregnant or breast-feeding.
9. Prior malignancies except resected basal cell carcinoma or treated cervical carcinoma in situ.
10. Disease modifying treatment prior to study enrollment, including but not limited to use of androgens, eltrombopag, romiplostim, or immune suppression. Note: Supportive care measures such as G-CSF, blood transfusion support and antibiotics are allowable

Ages: 0 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of this trial is time from randomization to treatment failure or death from any cause. | Randomization to 2 years post-randomization
  The median time to failure or death will be compared on the two arms using the log-rank test. Failure of IST is defined as the date that a second definitive therapy was recommended (BMT, second course of ATG) and failure of BMT defined as the date that a second definitive therapy was recommended (second BMT, course of ATG).

SECONDARY OUTCOMES:
Comparison of subjects with failure of IST or BMT before or at 2 years | Randomization to 2 years post-randomization
  The proportion of subjects with failure of IST or BMT before or at 2 years. Failure of IST is defined as initiation of a second definitive therapy (BMT, second course of ATG) and failure of BMT defined as initiation of a second definitive therapy (second BMT, course of ATG).
Comparison of subjects with inadequate counts at 2 years among those who have not died or failed treatment. | Randomization to 2 years post-randomization
  The proportion of subjects with inadequate counts at 2 years among those who have not failed therapy or died. Adequate counts are defined as: Absolute Neutrophil Count (ANC) >1 x 10^9/L, Hemoglobin >10g/dL, and Platelets >50 x10^9/L.
Comparison of subjects on immune suppression therapy at 2 years among those who have not died or failed treatment. | Randomization to 2 years post-randomization
  The proportion of subjects on immune suppression therapy at 2 years among those who have not failed therapy or died. Immune suppression is defined as systemic therapies necessary to treat SAA or GVHD (cyclosporine, tacrolimus, etc.). Isolated treatment with topical agents will not be considered as immune suppression therapy.
Estimate the time from randomization to initiation of IST or BMT. | Randomization through Day 100
  The median time in days from randomization to initiation of IST or BMT will be estimated. Initiation of therapy is first day of ATG for IST subjects, or day 0 (infusion day) for bone marrow transplant subjects.
Comparison of the frequency of failure to receive primary assigned therapy (IST or BMT) and reasons for the failure. | Randomization through Day 100
  The proportion of subjects who fail to receive randomized therapy and the frequency of reasons for failure.
Comparison of the incidence of bacteremia, viremia, and invasive fungal infection in the first two years after randomization in the IST and BMT arms. | Randomization through two years post randomization
  Proportion of subjects from the time of randomization in the first 2 years with each of the following:
  1. Documented bacteremia
  2. Documented viremia
  3. Documented invasive fungal infection (defined as confirmed or suspected fungal infection based upon imaging)
Estimate the median time to T- and B-cell immune reconstitution the first year for the URD BMT Arm | Initiation of therapy (Day 0) to 100 days, 180 days, 1 year and 2 years
  Absolute CD3, CD4, CD8, CD19, and CD56 (NK cell) numbers will be tracked at 100 days, 180 days, 1 year and 2 years post initiation of therapy in URT BMT arm. IgG levels free of IVIG replacement will be collected at the same timepoints. The median time to T- and B-cell reconstitution will be estimated.
Comparison of overall survival at 1 and 2 years from randomization in both arms. | Randomization to one year, randomization to two years
  Proportion of subjects who have died at 1 year and 2 years after randomization for any reason.
Comparison of treatment-related mortality (TRM) at 1 and 2 years from randomization in both arms. | Randomization to 1 year, randomization to 2 years
  Proportion of subjects who have died at 1 year and 2 years after randomization due to treatment-related reasons. TRM is defined as death in recipients without relapse or progression of their disease. Non-medical, accidental causes of death, e.g., natural disasters, are not considered TRM.
Comparison of the median time from randomization to and rates of neutrophil recovery on both arms | Randomization to 100 days, 180 days, 1 year and 2 years
  The time from randomization to neutrophil recovery. Neutrophil recovery is defined as ANC 0.5 x109/L for 3 consecutive measures for neutrophils (recovery date is the first date).
Comparison of the median time from randomization to and rate of platelet recovery on both arms | Randomization to 100 days, 180 days, 1 year and 2 years
  The time from randomization to platelet recovery. Platelet recovery is defined as platelet levels >= 20 x10^9/L for 3 consecutive measures (recovery is the first date) with no platelet transfusions for 1 full week.
Comparison of the median time from randomization to and rates of red blood cell recovery on both arms | Randomization to 100 days, 180 days, 1 year and 2 years
  The time from randomization to red blood cell recovery. Red blood cell recovery is defined as RBC hemoglobin level >= 8g/dL and 10g/dL with no RBC transfusions for 4 weeks.
Comparison of the median time from initiation of therapy to and rates of neutrophil recovery on both arms | Initiation of therapy to 100 days, 180 days, 1 year and 2 years
  The time from initiation of therapy (defined as Day 1 for patients randomized to IST and Day 0 for patients randomized to URD BMT) to neutrophil recovery. Neutrophil recovery is defined as ANC 0.5 x109/L for 3 consecutive measures for neutrophils (recovery date is the first date).
Comparison of the median time from initiation of therapy to and rate of platelet recovery on both arms | Initiation of therapy to 100 days, 180 days, 1 year and 2 years
  The time from initiation of therapy (defined as Day 1 for patients randomized to IST and Day 0 for patients randomized to URD BMT) to platelet recovery. Platelet recovery is defined as platelet levels >= 20 x10^9/L for 3 consecutive measures (recovery is the first date) with no platelet transfusions for 1 full week.
Comparison of the median time from initiation of therapy to and rates of red blood cell recovery on both arms. | Randomization to 100 days, 180 days, 1 year and 2 years
  The time from initiation of therapy (defined as Day 1 for patients randomized to IST and Day 0 for patients randomized to URD BMT) to red blood cell recovery. Red blood cell recovery is defined as RBC hemoglobin level >= 8g/dL and 10g/dL with no RBC transfusions for 4 weeks.
Estimate the rates of engraftment in patients who are randomized to URD BMT. | Randomization to 3-5 years
  Proportion of subjects with engraftment in patients who receive URD BMT.
Estimate the rates of primary graft failure in patients who are randomized to URD BMT . | Randomization to 3-5 years
  Proportion of subjects with primary graft failure in patients who receive URD BMT. Primary graft failure is defined as failure to achieve neutrophil recovery by Day +28 following a conditioning regimen induced neutrophil nadir < 0.5 x10^9/L.
Estimate the rates of secondary graft failure in patients who are randomized to URD BMT . | Randomization to 3-5 years
  Proportion of subjects with secondary graft failure in patients who receive URD BMT. Secondary graft failure will be defined as a fall in the neutrophil count after documented primary engraftment to < 0.5 x10^9/L sustained for more than three days that cannot be attributed to other causes such as drugs, infection, GVHD, etc., and is not responsive to G-CSF or GM-CSF.
Estimate the rates of grade II-IV acute GVHD in patients who are randomized to URD BMT . | Randomization to 3-5 years
  Proportion of subjects with grade II-IV in patients who receive URD BMT.
Estimate the rates of grade III-IV acute GVHD in patients who are randomized to URD BMT. | Randomization to 3-5 years
  Proportion of subjects with grade III-IV acute GVHD in patients who receive URD BMT.
Estimate the rates of severe chronic GVHD in patients who are randomized to URD BMT. | Randomization to 3-5 years
  Proportion of subjects with severe chronic GVHD in patients who receive URD BMT.
Estimate the rates of response of patients randomized to IST | Randomization to 100 days, 180 days, 1 year and 2 years
  Proportion of subjects with IST response. IST response criteria is:
  Complete Response: Hemoglobin ≥10 g/dL and ANC ≥1x10^9/L and Platelets ≥100x10^9/L Very Good Partial Response: Hemoglobin ≥8 g/dL and ANC ≥0.5x10^9/L and Platelets ≥50x10^9/L Partial Response: Hemoglobin ≥8 g/dL and ANC ≥0.5x10^9/L and Platelets ≥20x10^9/L and transfusion independent No Response (failure): Hemoglobin <8 g/dL or ANC <0.5x10^9/L or Platelets <20x10^9/L Lost Response: A lost response is captured by not meeting hematologic response criteria at a particular time point after having an initial response (complete, very good partial, or partial), or the need for additional treatment.
Estimate the rates of failure of patients randomized to IST | Randomization to 100 days, 180 days, 1 year and 2 years
  Proportion of subjects with IST failure at 6 months (defined as Hemoglobin <8 g/dL or ANC <0.5x10^9/L or Platelets <20x10^9/L).
Describe the secondary therapies given and outcomes achieved for patients failing initial therapy | Randomization to 3-5 years
  Collect secondary therapies given for failure of primary randomized therapy (BMT after IST, second course of IST, second BMT). For the outcome after subsequent therapy, the median survival time will be estimated.
Comparison of rates of secondary MDS, AML, other subsequent neoplasms, and development of Paroxysmal Nocturnal Hemoglobinuria in both treatment arms for the duration of the trial. | Randomization to 3-5 years
  Proportion of subjects in each treatment arm with i) subsequent neoplasms, ii) presence of a PNH clone at time of randomization who go on to develop symptomatic PNH through the duration of the protocol.
Comparison of HR-QoL score between patients randomized to both arms | Randomization to 2 years post-randomization, randomization to up to 5 years post-randomization
  Change in score between baseline and two years and the trajectory of change over all timepoints.
Comparison of gonadal function values between patients randomized to both arms | Randomization to 1 year post-randomization, randomization to 2 years post-randomization, and randomization to up to 5 years post-randomization
  Proportion of subjects with gonadal function values outside the expected percentile for that age.

CONTACTS AND LOCATIONS:
Overall Officials: David Williams, MD, Principal Investigator — Boston Children's Hospital; Michael Pulsipher, MD, Principal Investigator — University of Utah; Bronwen Shaw, MD, Principal Investigator — CIBMTR/Medical College of Wisconsin (MCW)
Locations (52):
- United States (50):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas, Little Rock, Arkansas
  - Loma Linda, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCLA, Los Angeles, California
  - Children's Hospital & Research Center Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Stanford, Palo Alto, California
  - Rady Children's Hospital San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Nemours Children's Hospital, Delaware, Wilmington, Delaware
  - Children's National Hospital, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Hospital of Atlanta/Emory, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University Hospital/Riley Hospital for Children, Indianapolis, Indiana
  - Children's Hospital NOLA, New Orleans, Louisiana
  - Maine Health, Scarborough, Maine
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Mayo Clinic Rochestser, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University in St. Louis, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Levine Children's Hospital, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Children's Medical Center Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Methodist Healthcare, San Antonio, Texas
  - University of Utah/Primary Children's Hospital, Salt Lake City, Utah
  - Children's Hospital of the King's Daughter, Norfolk, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Canada (2):
  - British Columbia Children's, Vancouver, British Columbia
  - Winnipeg CancerCare Manitoba, Winnipeg, Manitoba